CLINICAL TRIAL: NCT02359981
Title: MyBehavior: Persuasion by Adapting to User Behavior and User Preference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1302003617
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Weight Loss
Keywords: Weight loss, Fitness
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic suggestions (Active Comparator): Control group participants received suggestions generated by the a nutritionist and exercise trainer. These suggestions didn't relate to user's life or their past behavior.
  Interventions: Behavioral: Generic suggestions; Device: Smartphone
- MyBehavior (Experimental): Experiment group participants received personalized suggestions from MyBehavior that relates their life and past behavior.
  Interventions: Behavioral: MyBehavior; Device: Smartphone

INTERVENTIONS:
Behavioral: MyBehavior — The intervention automatically provides personalized suggestions based on users behavior and user context. Suggestions relates to users life and how often they have done them in the past. Since the suggestions relate to users' lives, they are easy to follow.
  Arms: MyBehavior
Behavioral: Generic suggestions — A nutritionist and an exercise trainer jointly created 45 food and exercise suggestions based on guidelines posted by the NIH. These suggestions ask users to walk for 30 minutes or eat healthier foods. These suggestions however doesn't personalize to users daily behavior into account.
  Arms: Generic suggestions
Device: Smartphone — An Android Smartphone with operating system version higher than 2.2

SUMMARY:
MyBehavior is a mobile application with a suggestion engine that learns a user's physical activity and dietary behavior, and provides finely-tuned personalized suggestions. To our knowledge, MyBehavior is the first smartphone app to provide personalized health suggestions automatically, going beyond commonly used one-size-fits-all prescriptive approaches, or tailored interventions from health-care professionals. MyBehavior uses an online multi-armed bandit model to automatically generate context-sensitive and personalized activity/food suggestions by learning the user's actual behavior. The app continually adapts its suggestions by exploiting the most frequent healthy behaviors, while sometimes exploring non-frequent behaviors, in order to maximize the user's chance of reaching a health goal (e.g. weight loss).

DETAILED DESCRIPTION:
A dramatic rise in self-tracking applications for smartphones has occurred recently. Rich user interfaces make manual logging of users' behavior easier and more pleasant; sensors make tracking effortless. To date, however, feedback technologies have been limited to providing counts or attractive visualization of tracked data. Human experts (health coaches) have needed to interpret the data and tailor make customized recommendations. No automated recommendation systems like Pandora, Netflix or personalized search for the web have been available to translate self-tracked data into actionable suggestions that promote healthier lifestyle without needing to involve a human interventionist.

MyBehavior aims to fill this gap. It takes a deeper look into physical activity and dietary intake data and reveal patterns of both healthy and unhealthy behavior that could be leveraged for personalized feedback. Based on common patterns from a user's life, suggestions are created that ask users to continue, change or avoid existing behaviors to achieve certain fitness goals. Such an approach is different from existing literature in two important aspects: (1) suggestions are contextualized to a user's life and are built on existing user behaviors. As a result, users can act on these suggestions easily, with minimal effort and interruption to daily routines; (2) unique suggestions are created for each individual. This personalized approach differs from traditional one-size-fits-all or targeted intervention models where identical suggestions are applied for groups of similar people or the entire population.

ELIGIBILITY:
Inclusion Criteria:

* In relatively healthy condition. Also, users must be interested in health and fitness.

Exclusion Criteria:

* Individuals with physical disability and dietary problems are excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
User intentions to follow automated suggestions and behavior change | 3 weeks
  The primary outcome is to measure efficacy of MyBehavior suggestions. Efficacy will be measured in two dimensions (1) whether users intend to follow the automated suggestions from MyBehavior (2) effectiveness of automated suggestions in actual behavior change.
  User intentions towards following MyBehavior suggestions are measured using a 5 point likert scale. The investigators will ask users to rate whether they can follow the suggestions on an average day within a scale of 1-5 (1- I can't follow the suggestion, 5 - I can easily follow the suggestion).
  On the other hand, behavior change is measured from food (calories in per meal consumed) and activity (walking, running or exercise durations per day etc.) log collected using their smartphone. Regarding physical activity, how much physical activity users are performing will be compared across experiment conditions. Similarly, calorie consumption change in food will be used to compare dietary behavior change.

SECONDARY OUTCOMES:
Usability improvements of automated suggestions | 3 weeks
  MyBehavior is the first system to provide health suggestions for food and activity automatically. Thus there are scopes of usability improvement on how to effectively present the automatically generated information to the user. Qualitative interviews at the end of study will be conducted to gather user experience of using MyBehavior. This interviews will help to build a better and more usable version of MyBehavior for future larger scale deployments.

CONTACTS AND LOCATIONS:
Overall Officials: Mashfiqui Rabbi, BS, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

REFERENCES:
- [Derived] Rabbi M, Pfammatter A, Zhang M, Spring B, Choudhury T. Automated personalized feedback for physical activity and dietary behavior change with mobile phones: a randomized controlled trial on adults. JMIR Mhealth Uhealth. 2015 May 14;3(2):e42. doi: 10.2196/mhealth.4160. PMID 25977197